CLINICAL TRIAL: NCT01628692
Title: A Phase 2, Open-Label Study of Daclatasvir (BMS-790052) and TMC435 in Combination With or Without Ribavirin (RBV) For Treatment-Naive Subjects or Null Responders to Prior Peginterferon Alfa (PegIFN)/RBV Therapy With Genotype 1 Chronic Hepatitis C
Brief Title: Study of Daclatasvir (BMS-790052) and Simeprevir (TMC435) in Patients With Genotype 1 Chronic Hepatitis C Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-062; 2012-000070-28 (EudraCT Number)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Simeprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: (Genotype 1b) Daclatasvir + Simeprevir (Experimental): Participants with hepatitis C virus genotype 1b received daclatasvir, 30 mg, once daily with or without food + simeprevir, 150 mg, once daily with a meal for 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Simeprevir
- Cohort 2: (Genotype 1b) Daclatasvir + Simeprevir + Ribavirin (Experimental): Participants with hepatitis C virus genotype 1b received daclatasvir, 30 mg, once daily with or without food + simeprivir, 150 mg, once daily with a meal + ribavirin, twice daily with food (patients weighing <75 kg received a total ribavirin dose of 1000 mg per day; those weighing >=75 kg received 1200 mg per day) for 12 weeks.
  Interventions: Drug: Daclatasvir; Drug: Simeprevir
- Cohort 3: (Genotype 1a) Daclatasvir + Simeprevir + Ribavirin (Experimental): Participants with hepatitis C virus genotype 1a received daclatasvir, 30 mg, once daily with or without food + simeprevir, 150 mg, once daily with a meal + ribavirin, twice daily with food (patients weighing <75 kg received a total ribavirin dose of 1000 mg per day; those weighing >=75 kg received 1200 mg per day) for 12 weeks.
  Interventions: Drug: Daclatasvir; Drug: Simeprevir; Drug: Ribavirin
- Cohort 4: (Genotype 1a) Daclatasvir + Simeprevir + Ribavirin (Experimental): Participants with hepatitis C virus genotype 1a received daclatasvir, 30 mg, once daily with or without food + simeprivir, 150 mg, once daily with a meal + ribavirin, twice daily with food (patients weighing <75 kg received a total ribavirin dose of 1000 mg per day; those weighing >=75 kg received 1200 mg per day.
  Interventions: Drug: Daclatasvir; Drug: Simeprevir; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Tablets, oral, 30 mg, once daily
  Other Names: BMS-790052
Drug: Simeprevir — Capsule, oral, 150 mg, once daily
  Other Names: TMC435
Drug: Ribavirin — Tablets, oral, 500-600 mg, twice daily
  Arms: Cohort 3: (Genotype 1a) Daclatasvir + Simeprevir + Ribavirin; Cohort 4: (Genotype 1a) Daclatasvir + Simeprevir + Ribavirin

SUMMARY:
The purpose of this study is to assess the safety and efficacy of daclatasvir and simeprevir with and without ribavirin for genotype 1 chronic hepatitis C virus infection in patients who are treatment-naive or null responders to previous pegylated interferon/ribavirin therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Hepatitis C virus (HCV) genotype 1a or 1b
* Males and females, ≥18 years of age
* HCV RNA ≥10,000 IU/mL
* Participants with compensated cirrhosis are permitted

  * Advanced fibrosis (F3/F4) is capped at approximately 35% of the total treated population with a minimum of 20% F4 patients
  * If no cirrhosis, a liver biopsy within 3 years prior to enrollment
  * If cirrhosis is present, any prior liver biopsy

Key Exclusion Criteria:

* Liver or any other transplant (other than cornea and hair)
* Evidence of a medical condition contributing to chronic liver disease other than HCV infection
* Current or known history of cancer, (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment
* Evidence of decompensated liver disease including, but not limited to, radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
* Patients infected with HIV or hepatitis B virus
* Gastrointestinal disease impacting absorption of study drug
* Uncontrolled diabetes or hypertension
* Prior exposure to an HCV direct-acting agent
* Any criteria that would exclude the patient from receiving ribavirin
* Absolute neutrophil count <1.5*1,000,000,000 cells/L (<1.2*1,000,000,000 cells/L for Black/African Americans)
* Platelets <90*1,000,000,000 cells/L
* Hemoglobin <12 g/dL for females, <13 g/dL for males
* Alanine aminotransferase ≥5*upper limit of normal
* In patients without cirrhosis, total bilirubin ≥2 mg/dL unless patient has a documented history of Gilbert's disease
* In patients with cirrhosis, total bilirubin o ≥1.5 mg/dL
* International normalized ratio ≥1.7
* QTcF or QTcB >500 mSec
* Creatinine clearance ≤50 mL/min
* Alpha fetoprotein (AFP) >100 ng/mL OR
* AFP ≥50 ng/mL and ≤100 ng/mL requiring liver ultrasound
* Albumin <3.5 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (7):
  - San Francisco General Hospital, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Lutherville, Maryland
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Texas Clinical Research Institute, Llc, Arlington, Texas
  - Metropolitan Research, Fairfax, Virginia
- Local Institution, Buenos Aires, Buenos Aires, Argentina
- France (6):
  - Local Institution, Créteil
  - Local Institution, Limoges
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Gyula
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia

REFERENCES:
- [Derived] Zeuzem S, Hezode C, Bronowicki JP, Loustaud-Ratti V, Gea F, Buti M, Olveira A, Banyai T, Al-Assi MT, Petersen J, Thabut D, Gadano A, Pruitt R, Makara M, Bourliere M, Pol S, Beumont-Mauviel M, Ouwerkerk-Mahadevan S, Picchio G, Bifano M, McPhee F, Boparai N, Cheung K, Hughes EA, Noviello S; LEAGUE-1 Study Team. Daclatasvir plus simeprevir with or without ribavirin for the treatment of chronic hepatitis C virus genotype 1 infection. J Hepatol. 2016 Feb;64(2):292-300. doi: 10.1016/j.jhep.2015.09.024. Epub 2015 Oct 8. PMID 26453968
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 centers in 6 countries.
Pre-assignment Details: Of the 230 participants enrolled, 168 received treatment.
Groups:
- Genotype 1b: Daclatasvir + Simeprevir (Naive): Participants with no prior treatment of hepatitis C virus genotype 1b. Received daclatasvir 30 mg with or without food and simeprevir 150 mg with a light to standard meal once daily (QD), for a period of 12 weeks or 24 weeks based on re-randomization and continued into a post-treatment follow-up period.
- Genotype 1b: Daclatasvir + Simeprevir (Null): Participants with hepatitis C virus genotype 1b, and who never attained ≥2 log10 decline in hepatitis C virus RNA levels after at least 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food and simeprevir 150 mg with a light to standard meal QD, for a period of 12 or 24 weeks based on re-randomization and continued into post-treatment follow-up.
- Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive): Participants with no prior treatment of hepatitis C virus genotype 1b. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>= 75 kg, respectively) ribavirin twice daily (BID) for a period of 12 or 24 weeks based on re-randomization and continued into post-treatment follow-up.
- Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null): Participants with hepatitis C virus genotype 1b, who never attained ≥2 log10 decline in hepatitis C virus RNA level after 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>=75 kg, respectively) ribavirin BID were continued to receive treatment for a period of 12 or 24 weeks based on re-randomization and continued into post-treatment follow-up period.
- Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive): Participants with no prior treatment of hepatitis C virus genotype 1a. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>=75 kg, respectively) ribavirin BID for a period of 24 weeks and continued into post-treatment follow-up period of 24 weeks.
- Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null): Participants with hepatitis C virus genotype 1a, who never attained ≥2 log10 decline in hepatitis C virus genotype RNA level after 12 weeks of prior therapy. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>=75 kg, respectively) ribavirin BID for a period of 24 weeks and continued into post-treatment follow-up period of 24 weeks.
Period: Overall Study
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Started | 53 | 23 | 51 | 20 | 12 | 9
Completed | 46 | 17 | 43 | 19 | 8 | 0
Not Completed | 7 | 6 | 8 | 1 | 4 | 9
Not completed — Lack of Efficacy | 4 | 4 | 5 | 1 | 4 | 7
Not completed — Adverse Event | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Poor compliance/noncompliance | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Completed 12 Week only | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on the treated participants defined as all randomized participants who received at least 1 dose of active study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null) | Total
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9 | 168
Age, Customized [Number; unit: participants]
  <21 years | 0 | 0 | 0 | 1 | 1 | 0 | 2
  21-<65 years | 41 | 19 | 42 | 11 | 11 | 9 | 133
  >=65 years | 12 | 4 | 9 | 8 | 0 | 0 | 33
Gender [Count of Participants; unit: Participants]
  Female | 31 | 11 | 26 | 11 | 5 | 2 | 86
  Male | 22 | 12 | 25 | 9 | 7 | 7 | 82
Hepatitis C Virus RNA Distribution [Number; unit: participants]
  <800,000 IU/mL | 12 | 3 | 11 | 4 | 5 | 0 | 35
  ≥800,000 IU/mL | 41 | 20 | 40 | 16 | 7 | 9 | 133
Randomization Stratum [Number; unit: participants]
  Hepatitis C Virus Genotype 1b | 53 | 23 | 51 | 20 | 0 | 0 | 147
  Hepatitis C Virus Genotype 1a | 0 | 0 | 0 | 0 | 12 | 9 | 21

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Week 4
Description: RVR was defined as hepatitis C virus (HCV) RNA levels to be <lower limit of quantitation, target not detected at Week 4. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4
Population: All treated participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants | 79.2 [72.1 to 86.4] | 69.6 [57.3 to 81.9] | 68.6 [60.3 to 77.0] | 85 [74.8 to 95.2] | 75 [59.0 to 91.0] | 33.3 [13.2 to 53.5]

2. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as hepatitis C virus (HCV) RNA levels to be <lower limit of quantitation, target not detected at Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12
Population: All treated participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Groups:
- Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null): Participants with no prior treatment of hepatitis C virus genotype 1b. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>= 75 kg, respectively) ribavirin twice daily (BID) for a period of 12 or 24 weeks based on re-randomization and continued into post-treatment follow-up.
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants | 84.9 [78.6 to 91.2] | 73.9 [62.2 to 85.6] | 82.4 [75.5 to 89.2] | 90 [81.4 to 98.6] | 66.7 [49.2 to 84.1] | 11.1 [0 to 24.5]

3. Primary Outcome: Percentage of Participants With Sustained Virologic Response Rate at Post-treatment Week 12 (SVR12)
Description: SVR12 rate was defined as hepatitis C virus (HCV) RNA levels to be <lower limit of quantitation, target detected or target not detected, at post-treatment Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Post Treatment Week 12 (Follow-up period)
Population: All participants who were randomized and received at least 1 dose of active study therapy (daclatasvir, simeprevir, ribavirin).
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants | 84.9 [78.6 to 91.2] | 69.6 [57.3 to 81.9] | 74.5 [66.7 to 82.3] | 95 [88.8 to 100] | 66.7 [49.2 to 84.1] | 0 [NA to NA] — As none of the participants responded to SVR12, 80% confidence interval value is not available.

4. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR were defined as hepatitis C virus (HCV) RNA levels to be <lower limit of quantitation, target not detected at both Week 4 and Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4 and Week 12
Population: All treated participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants | 71.7 [63.8 to 79.6] | 60.9 [47.8 to 73.9] | 62.7 [54.1 to 71.4] | 75 [62.6 to 87.4] | 58.3 [40.1 to 76.6] | 11.1 [0 to 24.5]

5. Secondary Outcome: Percentage of Participants With End of Treatment Response (EOTR)
Description: EOTR were defined as hepatitis C virus (HCV) RNA levels <lower limit of quantitation, target not detected at end of treatment. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: End of treatment (Week 24)
Population: All treated participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants | 88.7 [83.1 to 94.3] | 78.3 [67.2 to 89.3] | 78.4 [71.1 to 85.8] | 95 [88.8 to 100] | 66.7 [49.2 to 84.1] | 0 [NA to NA] — As none of the participants responded at EOT, hence 80% confidence interval value is not available.

6. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Week 12 (SVR12) by rs12979860 Single Nucleotide Polymorphisms in the IL-28B Gene Categories
Description: Participants were categorized into 3 genotypes based on single nucleotide polymorphisms in the IL28B gene. SVR12 was defined as hepatitis C virus (HCV) RNA levels below lower limit of quantitation, target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Baseline, post-treatment Week 12 (Follow-up period)
Population: All treated participants. Here 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive) | Genotype 1b: Daclatasvir + Simeprevir (Null) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1b: Daclatasvir + Simeprevir + Ribavirin (Null) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Naive) | Genotype 1a: Daclatasvir + Simeprevir + Ribavirin (Null)
Number analyzed (Participants) | 53 | 23 | 51 | 20 | 12 | 9
Percentage of participants
  IL28B Genotype CC type (n= 16,1,13,1,3,0) | 87.5 | 100 | 84.6 | 100 | 66.7 | NA — As no participant was evaluable for assessment, hence value is not available.
  IL28B Genotype CT type (n= 22,15, 28,10,9,8) | 95.5 | 60 | 82.1 | 90 | 66.7 | 0
  IL28B Genotype TT type (n= 12,6,10,7,0,1) | 66.7 | 83.3 | 40 | 100 | NA — No participants were available for assessment | 0

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Discontinuations Due to Adverse Events (AEs) and Who Died
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Based on the severity, AEs were categorized as Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: From start of treatment (Day 1) up to 7 days post last dose of study treatment (Week 24)
Population: All treated participants.
Measure: Number; unit: Participants
Groups:
- Genotype 1b: Daclatasvir + Simeprevir (Naive + Null): Participants with and without prior treatment of hepatitis C virus genotype 1b and who never attained ≥2 log10 decline in hepatitis C virus RNA levels after at least 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food and simeprevir 150 mg with a light to standard meal once daily (QD), for a period of 12 weeks or 24 weeks based on re-randomization and continued into a post-treatment follow-up period.
- Genotype1b: Daclatasvir +Simeprevir + Ribavirin (Naive + Null): Participants with and without prior treatment of hepatitis C virus genotype 1b and who never attained ≥2 log10 decline in hepatitis C virus RNA levels after at least 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>= 75 kg, respectively) ribavirin twice daily (BID) for a period of 12 or 24 weeks based on re-randomization and continued into post-treatment follow-up.
- Genotype1a: Daclatasvir +Simeprevir + Ribavirin(Naive + Null): Participants with and without prior treatment of hepatitis C virus genotype 1a and who never attained ≥2 log10 decline in hepatitis C virus RNA levels after at least 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>=75 kg, respectively) ribavirin BID for a period of 24 weeks and continued into post-treatment follow-up period of 24 weeks.
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive + Null) | Genotype1b: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) | Genotype1a: Daclatasvir +Simeprevir + Ribavirin(Naive + Null)
Number analyzed (Participants) | 76 | 71 | 21
Participants
  SAEs | 7 | 3 | 1
  AEs Leading to Discontinuation | 2 | 2 | 0
  Death | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment (Day 1) up to 7 days post last dose of study treatment (Week 24)
Description: On-Treatment Period
Groups:
- Genotype1a: Daclatasvir +Simeprevir + Ribavirin (Naive + Null): Participants with and without prior treatment of hepatitis C virus genotype 1a and who never attained ≥2 log10 decline in hepatitis C virus RNA levels after at least 12 weeks of prior therapy with peginterferon/ribavirin. Received daclatasvir 30 mg with or without food, simeprevir 150 mg with a light to standard meal QD, and weight stratified (1000/1200 mg for participants weighing <75/>=75 kg, respectively) ribavirin BID for a period of 24 weeks and continued into post-treatment follow-up period of 24 weeks.
Arm/Group | Genotype 1b: Daclatasvir + Simeprevir (Naive + Null) | Genotype1b: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) | Genotype1a: Daclatasvir +Simeprevir + Ribavirin (Naive + Null)
Serious Adverse Events (participants affected / at risk) | 7/76 | 3/71 | 1/21
Other Adverse Events (participants affected / at risk) | 49/76 | 63/71 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 1b: Daclatasvir + Simeprevir (Naive + Null) (N=76) | Genotype1b: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) (N=71) | Genotype1a: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) (N=21)
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 1b: Daclatasvir + Simeprevir (Naive + Null) (N=76) | Genotype1b: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) (N=71) | Genotype1a: Daclatasvir +Simeprevir + Ribavirin (Naive + Null) (N=21)
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 12 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 5 | 4
Hot flush (Vascular disorders) | 0 | 1 | 2
Irritability (General disorders) | 3 | 1 | 2
Sleep disorder (Psychiatric disorders) | 5 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 5
Depressed mood (Psychiatric disorders) | 0 | 0 | 2
Fatigue (General disorders) | 6 | 11 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 12 | 3
Insomnia (Psychiatric disorders) | 4 | 7 | 1
Nausea (Gastrointestinal disorders) | 14 | 11 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 15 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 10 | 9 | 2
Asthenia (General disorders) | 15 | 16 | 5
Dry eye (Eye disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 16 | 10 | 6
Hypertension (Vascular disorders) | 5 | 2 | 1
Disturbance in attention (Nervous system disorders) | 2 | 0 | 2
Influenza like illness (General disorders) | 5 | 1 | 3
Jaundice (Hepatobiliary disorders) | 1 | 4 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 9 | 3
Visual acuity reduced (Eye disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 0
Chills (General disorders) | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 6 | 5 | 4
Pain (General disorders) | 3 | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.